CLINICAL TRIAL: NCT00957775
Title: Computer-delivered Psychosocial Intervention for Adolescent Substance Use Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Development and Research Institutes, Inc. (Other)
Collaborators: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Lisa A. Marsch, Ph.D., National Development and Research Institutes, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA025072 (NIH); R01DA025072 (NIH)
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2009-08-12 (Estimated); Status verified 2009-08

CONDITIONS: Substance-Related Disorders; Alcohol-Related Disorders; Marijuana Abuse
Keywords: Substance Abuse Treatment; Adolescents; Substance-Related Disorders; Alcohol-Related Disorders; Marijuana Abuse
MeSH Terms: conditions — Substance-Related Disorders; Alcohol-Related Disorders; Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): Participants will receive the usual care (e.g., individual therapy, group therapy, self-help groups) provided at the treatment site.
  Interventions: Behavioral: Usual care
- Computer-delivered ACRA (Experimental): Participants and willing caregivers will receive a computer-delivered intervention for 12 weeks, based on the Adolescent Community Reinforcement Approach to substance abuse treatment.
  Interventions: Behavioral: Computer-delivered ACRA

INTERVENTIONS:
Behavioral: Usual care — Participants will receive the usual care (e.g., individual therapy, group therapy, family therapy, self-help groups) provided at the treatment site.
  Other Names: treatment-as-usual (TAU)
  Arms: Usual care
Behavioral: Computer-delivered ACRA — Participants and willing caregivers will receive a computer-delivered intervention for 12 weeks, based on the Adolescent Community Reinforcement Approach to substance abuse treatment.
  Arms: Computer-delivered ACRA

SUMMARY:
The purpose of this study is to develop and evaluate the acceptability and preliminary efficacy of a web-based, skills training program for adolescents with substance use disorders.

DETAILED DESCRIPTION:
Substance use among youth remains a major public health problem. About half of all 12th graders have tried an illicit drug and over 72% of this same age group have used alcohol. Rates of abuse of prescription opioids among youth are estimated to have increased about 542% in the past decade. Although effective substance abuse treatment programs for youth exist, they are currently of limited reach. Only 1 in 10 adolescents who need substance abuse treatment receive any care. An interactive, computer-delivered psychosocial (skills-training) intervention has the potential to address these challenges, as it allows for complex interventions to be delivered at a low cost, without increasing demands on staff time or training needs. It may also be highly acceptable to youth and enable widespread dissemination of science-based treatment in a manner that ensures fidelity.

In this project, we plan to develop and evaluate the acceptability and preliminary efficacy of a web-based, skills training program for adolescents with substance use disorders. The content of this program will be based in a model of psychosocial substance abuse treatment for youth that has been shown to be effective in prior scientific research. It will be provided via an interactive, delivery system that employs informational technologies that are effective in promoting relevant knowledge and skills. Adolescents in substance abuse treatment will help shape the development of this program. To our knowledge, the planned program will be the first interactive program to provide comprehensive, psychosocial substance abuse treatment to adolescents via computer-based technology.

This research will contribute new information relevant to increasing the delivery of science-based psychosocial treatment to adolescents with substance use disorders in a manner that is cost-effective and which may promote the adoption of effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of non-nicotine alcohol or drug use disorder
* English speaking
* Parental consent to participate for adolescents under the age of 18.

Exclusion Criteria:

* Clinical diagnosis of psychiatric disorders that require intensive level of services, such as active psychosis, active mania or active suicidality
* Plan to move out of the area within the next 3 months
* Insufficient ability to understand and provide informed consent/assent to participate
* Lack sufficient ability to use English to participate in the consent/assent process, the interventions or assessments

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
substance use | 16 weeks
acceptability of intervention | 12 weeks

SECONDARY OUTCOMES:
HIV risk behavior | 16 weeks
psychosocial functioning | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Marsch, Ph.D., Principal Investigator — National Development and Research Institutes, Inc.
Locations (1):
- National Development and Research Institutes, Inc.; St. Luke's-Roosevelt Hospital Center, New York, New York, United States